CLINICAL TRIAL: NCT00352469
Title: 12 Week Prospective Double Blind Placebo Controlled Randomized Trial of Seroquel SR for Alcohol Dependence and Comorbid Anxiety
Brief Title: Trial of Seroquel SR for Alcohol Dependence and Comorbid Anxiety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: S. Pirzada Sattar, M.D., Assistant Professor, Creighton University Department of Psychiatry
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRUSQUET408
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Alcoholism; Anxiety Disorders; Generalized Anxiety Disorder; Post-Traumatic Stress Disorder; Panic Disorder; Obsessive-Compulsive Disorder
Keywords: Alcoholism; Anxiety; GAD; PTSD; Panic Disorder; OCD
MeSH Terms: conditions — Alcoholism; Anxiety Disorders; Generalized Anxiety Disorder; Stress Disorders, Post-Traumatic; Panic Disorder; Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Placebo Comparator): Subjects will be randomized to receive either Seroquel SR or placebo
  Interventions: Drug: Seroquel XR

INTERVENTIONS:
Drug: Seroquel XR — Day 1 and 2 Seroquel XR 50 mg; Day 3-4 Seroquel XR 150mg;Day 5-42 Seroquel XR 300-400mg

SUMMARY:
Alcohol use disorders (AUDs) are a major problem facing our society. Their treatment is complex, and involves multiple behavioral and pharmacotherapy interventions. There are 3 approved medications for AUDs, but their efficacy for AUDs that co-exist with anxiety disorders is unknown. This study explores the effects of the medication, sustained-release quetiapine fumarate (Seroquel SR) for the treatment of alcohol dependence and co-morbid anxiety. Primary outcome measure is the amount of alcohol used. Secondary outcome measures include craving for alcohol, length of sobriety from drinking and level of anxiety with Seroquel SR.

DETAILED DESCRIPTION:
STUDY OBJECTIVES:

The objective of this proposal is to study the efficacy of the medication Seroquel SR for the treatment of alcohol dependence and co-morbid anxiety in a prospective double blind placebo-controlled randomized clinical study. Patients, meeting the DSM-IV criteria for Alcohol Dependence and an Anxiety Disorder, will be enrolled and randomized to receive placebo or Seroquel SR. All subjects will be referred to usual treatment program, where they can receive group/self help group therapy.

Method:

This is a 12-week prospective, double blind placebo-controlled randomized clinical trial of Seroquel SR in patients who meet the Diagnostic and Statistical Manual of Psychiatric Disorders (DSM-IV) criteria for alcohol dependence and anxiety disorders. Potential candidates will be allowed sufficient time to review the consent document and ask questions about the trial prior to signing the consent document. Consenting adults will be randomized to receive active medication, Seroquel SR or placebo for 12-weeks. The study will enroll 20 patients, 10 will be randomized to receive Seroquel SR, and 10 will receive placebo. All participants will also be referred to usual alcohol treatment, including individual, group and/or self help group therapy (Alcoholics Anonymous).

Subjects will be randomized to receive either Seroquel SR or placebo. Dosing of Seroquel SR will occur on the following schedule: At the baseline visit, Seroquel SR will be started at 50 mg QHS for Day 1 and 2, and dose increase to 150 mg QHS on day 3-4, and increased further to 300 mg QHS from day 5-day 42. After day 5, the Seroquel SR dosage can be increased by up to 100 mg per week to a maximal dose of 400 mg per day. During the treatment period, dose reductions (because of physical illness or adverse event) are allowed for patients taking at least 200 mg per day.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of alcohol dependence and an anxiety disorder (generalized anxiety disorder, post traumatic disorder, panic disorder, obsessive compulsive disorder, etc.) based on Mini-International Neuropsychiatric Interview (MINI) for DSM IV.
2. Subject reports a minimum of 48 standard alcoholic drinks (or an average of 12 drinks/wk) in a consecutive 30-day period (i.e., a minimum of 40% days drinking), and has 2 or more days of heavy drinking (defined as ≥5 drinks/day in males and ≥4 drinks/day in females) in this same period as measured by the Time Line Follow Back.
3. Male and female patients between 19-65 years of age.
4. Ability to provide informed consent.
5. Medically and psychiatrically stable defined as not requiring inpatient treatment.

Exclusion Criteria:

1. Inability to provide informed consent.
2. Need for inpatient treatment
3. Need for inpatient detoxification for substance other than alcohol
4. Evidence of active dependence on a substance other than alcohol (with the exception of nicotine) as assessed by a urine drug screen.
5. Medically or psychiatrically unstable patients, defined as requiring inpatient treatment.
6. Pregnancy, nursing or refusal to use a reliable method of birth control in women.
7. Current treatment with other antipsychotic medications, which cannot be switched to Seroquel SR.
8. Patients with known allergy to Seroquel IR/SR or treatment failure to Seroquel IR/SR.
9. Exclude patients (pts) with unstable diabetes.
10. Exclude pts over 65
11. Exclude pts with dementia

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Aim 1: To determine whether Seroquel SR reduces alcohol use and prolongs sobriety as measured by the Time Line Follow Back Method and breathalyzer test in individuals with alcohol dependence and co-morbid anxiety. | Two Years

SECONDARY OUTCOMES:
Aim 2: To determine whether Seroquel SR decreases craving as measured by the Pennsylvania Craving Scale, in individuals with alcohol dependence and co-morbid anxiety. | Two Years
Aim 3: To determine whether Seroquel SR reduces anxiety symptoms as measured by the Hamilton Rating Scale for Anxiety (HAM-A), in individuals with alcohol dependence and co-morbid anxiety. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Pirzada Sattar, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Department of Psychiatry, Omaha, Nebraska, United States